CLINICAL TRIAL: NCT05634486
Title: Efficacy Study of the Multidisciplinary Therapeutic Approach to the Quality of Life of Patients With Functional Movement Disorders and Their Caregivers
Brief Title: Efficacy of the Multidisciplinary Treatment to the Quality of Life of With Functional Movement Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Fundación Caser (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1633-N-21
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Functional Neurological Disorder; Functional Movement Disorder
MeSH Terms: conditions — Conversion Disorder | interventions — Physical Therapy Modalities; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: 40 patients with functional movement disorders will be randomized into two arms of treatments: a one-month multidisciplinary treatment (physiotherapy + cognitive-behavioral therapy) versus a one-month psychoeducation sham intervention (control group).
Who Masked: Investigator
Masking Description: Movement disorders specialists will review the severity of symptoms as blinded raters in the 3th-month and 5th-month follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary therapeutic approach (Experimental): * Diagnosis of Functional Movement Disorders by one of the PI (Movement Disorders Specialist).
  * 12 physiotherapy sessions during one month (three 60-minute sessions per week) administered by a physiotherapist with experience in functional neurological disorders.
  * 4 cognitive-behavioral therapy sessions during one month (one 60-minute intervention per week) administered by a psychologist with experience in cognitive-behavioral therapy.
  Interventions: Behavioral: Multidisciplinary therapeutic approach (physiotherapy plus cognitive-behavioral therapy)
- Psychoeducation (Sham Comparator): * Diagnosis of Functional Movement Disorders by one of the PI (Movement Disorders Specialist).
  * 4 psychoeducational sessions (one 60-minute intervention per week) administered by a psychologist with experience in cognitive-behavioral therapy.
  Interventions: Other: Psychoeducation (Sham intervention)

INTERVENTIONS:
Behavioral: Multidisciplinary therapeutic approach (physiotherapy plus cognitive-behavioral therapy) — Patients randomly allocated to this arm of intervention will receive an ambulatory therapy regime of twelve 60-minute physiotherapy sessions plus four 60-minute psychotherapy sessions throughout one month of treatment
  Arms: Multidisciplinary therapeutic approach
Other: Psychoeducation (Sham intervention) — Patients randomly allocated to this arm of intervention will receive an ambulatory regime of four 60-minute non-organized psychoeducational sessions throughout one month of treatment.
  Arms: Psychoeducation

SUMMARY:
Randomized-clinical trial of multidisciplinary approach versus psychoeducation in patients with functional movement disorders: impact to their quality of life and their caregivers' quality of life. Patients with functional movement disorders are randomized in two arms of a one-month treatment (physiotherapy + cognitive-behavioral therapy versus psychoeducational as sham intervention) with a 3-month and 5-month follow-up where the investigators will measure the change in the patients' and caregivers' quality of life. Movement disorders specialists will review the severity of symptoms as blinded raters in the 3th-month and 5th-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Functional Movement Disorders (Espay and Lang, 2015)
* Patients should be 18 years old or older and capable of giving consent to freely and willingly participate in the study.
* Patients should be able to attend the one-month ambulatory regime and follow-up visits.

Exclusion Criteria:

* Any condition that avoid the patient from giving free consent to participate in the study.
* Any non-controlled psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life in patients with functional movement disorders measured by The 5-level EQ-5D version (EQ-5D-5L) - EQ visual analogue scale | 3th-month and 5th-month follow-ups
  Change in the patients' quality of life measured by changes in EQ-5D-5L - the EQ visual analogue scale (EQ VAS).
Quality of Life in patients with functional movement disorders measured by The 5-level EQ-5D version (EQ-5D-5L) - EQ-5D descriptive system. | 3th-month and 5th-month follow-ups
  Change in the patients' quality of life measured by changes in EQ-5D-5L - EQ-5D descriptive system. The digits for the five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) can be combined into a 5-digit number that describes the patient's health state.
Quality of Life in patients with functional movement disorders measured by the 36-Item Short Form Health Survey (SF-36) | 3th-month and 5th-month follow-ups
  Change in the patients' quality of life measured by changes in SF-36

SECONDARY OUTCOMES:
Quality of Life in caregivers of patients with functional movement disorders | 3th-month and 5th-month follow-ups
  Change in the caregivers' quality of life measured by changes in the Zarit Caregiver Burden Interview
Severity of functional neurological symptoms of patients with functional movement disorders measured by Clinical Global Impressions (CGI) Scale | 3th-month and 5th-month follow-ups
  Change in the patients' symptoms severity measured by changes in the Clinical Global Impressions (CGI) Scale - Severity
Improvement of functional neurological symptoms of patients with functional movement disorders | 3th-month and 5th-month follow-ups
  Improvement of the patients' symptoms severity measured by the Clinical Global Impressions (CGI) Scale - Improvement
Severity of functional neurological symptoms of patients with functional movement disorders | 3th-month and 5th-month follow-ups
  Change in the patients' symptoms severity measured by changes in the simplified-Functional Movement Disorders Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Mir, MD, PhD, Principal Investigator — Hospital Universitario Virgen del Rocío / Instituto de Biomedicina de Sevilla (IBiS)
Locations (1):
- Hospital Universitario Virgen del Rocío / Instituto de Biomedicina de Sevilla (IBiS), Seville, Spain

REFERENCES:
- [Derived] Macias-Garcia D, Mendez-Del Barrio M, Canal-Rivero M, Munoz-Delgado L, Adarmes-Gomez A, Jesus S, Ojeda-Lepe E, Carrillo-Garcia F, Palomar FJ, Gomez-Campos FJ, Martin-Rodriguez JF, Crespo-Facorro B, Ruiz-Veguilla M, Mir P. Combined Physiotherapy and Cognitive Behavioral Therapy for Functional Movement Disorders: A Randomized Clinical Trial. JAMA Neurol. 2024 Sep 1;81(9):966-976. doi: 10.1001/jamaneurol.2024.2393. PMID 39102249
- See also: Sponsor official statement of financial support — https://www.fundacioncaser.org/actividades/ayudas-investigacion-sociosanitaria/ayudas-la-investigacion-sociosanitaria-2021